CLINICAL TRIAL: NCT07128576
Title: A Multicenter Phase II Clinical Study of Romiplostim N01 for the Treatment of Thrombocytopenia Associated With Radiotherapy-Combined Treatment Regimens in Patients With Solid Tumors
Brief Title: Romiplostim N01 for the Treatment of Thrombocytopenia Associated With Radiotherapy-Combined Treatment Regimens in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, bujunguo, Doctor, Zhujiang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-078-01
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A: PLT 10-50×10^9/L romiplostim N01 (Experimental)
  Interventions: Drug: Romiplostim N01
- arm B: PLT 50-70×10^9/L romiplostim N01 (Experimental)
  Interventions: Drug: Romiplostim N01

INTERVENTIONS:
Drug: Romiplostim N01 — Romiplostim N01: 3-10 μg/kg(Initial dose 3 μ g/kg), qw, H.

SUMMARY:
With the development of modern medicine, targeted and immunotherapies have been widely adopted in clinical practice. Beyond conventional chemotherapy combination regimens, the integration of radiotherapy into multimodal treatment strategies has also expanded significantly.

While robust evidence supports the use of romiplostim for managing chemotherapy-induced thrombocytopenia (CIT), there is currently no clinical research evaluating its efficacy in treating thrombocytopenia associated with radiotherapy-combined treatment regimens in solid tumors.

To address this unmet clinical need, this study aims to evaluate the safety and efficacy of romiplostim N01 for injection in the treatment of radiotherapy-combined regimen-induced thrombocytopenia in solid tumor patients. The findings will establish evidence-based management strategies to optimize clinical decision-making in this context.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, regardless of gender; Histopathologically confirmed solid tumor patients (including but not limited to nasopharyngeal carcinoma, lung cancer, breast cancer, etc.);
* Prior radiotherapy (RT) ≥45Gy (including standalone RT, concurrent/sequential chemoradiotherapy, or RT combined with other antitumor therapies, with treatment duration ≥2 weeks), regardless of prior induction/adjuvant chemotherapy;
* Platelet count <75×10⁹/L within 3 days prior to enrollment, occurring during RT or within 1 month post-RT;
* Estimated survival ≥12 weeks at screening;
* ECOG score 0, 1, or 2;
* Premenopausal women/men of childbearing potential must agree to contraceptive measures during and for 6 months post-study; non-lactating patients;
* No participation in other drug clinical trials within 4 weeks prior to enrollment;
* Voluntary signing of informed consent after full comprehension of study requirements.

Exclusion Criteria:

* Patients with hematologic diseases, including lymphoma, leukemia, aplastic anemia, primary immune thrombocytopenia (ITP), myeloproliferative disorders, multiple myeloma, or myelodysplastic syndromes;
* Patients who experienced thrombocytopenia within 6 months prior to screening due to non-cancer treatments, including but not limited to EDTA-dependent pseudo-thrombocytopenia, hypersplenism, infection, or bleeding.
* Patients with brain tumors, brain metastases, bone marrow invasion, or bone marrow metastases;
* Patients with hemoglobin <50 g/L after red blood cell transfusion or erythropoietin (EPO) treatment, or absolute neutrophil count <1.0×10⁹/L after granulocyte colony-stimulating factor (G-CSF) treatment;
* Patients who experienced any arterial or venous thrombosis within 6 months prior to screening;
* Patients with severe cardiovascular diseases within 6 months prior to screening (e.g., NYHA Class III-IV heart failure), high-risk arrhythmias (e.g., atrial fibrillation), coronary stent placement, angioplasty, or coronary artery bypass grafting;
* Patients who received platelet transfusion within 5 days prior to enrollment;
* Patients who received thrombopoietin receptor agonist treatment within 4 weeks prior to study drug administration, recombinant human thrombopoietin (rhTPO) or rhIL-11 within 4 weeks prior to enrollment, or other platelet-enhancing traditional Chinese medicine within 1 week prior to enrollment;
* Patients with positive hepatitis C antibody and detectable HCV-RNA, positive hepatitis B surface antigen and detectable HBV-DNA, severe cirrhosis, HIV antibody positivity, or syphilis antibody positivity;
* Patients with ALT and AST ≥3×ULN (for subjects without liver metastasis) or ≥5×ULN (for subjects with liver metastasis) during screening;
* Patients with serum creatinine ≥1.5×ULN or estimated glomerular filtration rate (eGFR) ≤60 mL/min;
* Patients with known allergies or intolerances to the active ingredients or excipients of romiplostim N01 for injection;
* Patients who are pregnant, planning pregnancy, or breastfeeding;
* Patients deemed unsuitable for participation in the trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving ≥50×10⁹/L increase in platelet count (PLT) from baseline within 2 weeks | 2 weeks

SECONDARY OUTCOMES:
Proportion of patients achieving ≥50×10⁹/L increase in PLT from baseline within 4 weeks | 4 weeks
Time to first PLT recovery ≥100×10⁹/L | 1 month
Proportion of patients requiring platelet transfusions due to thrombocytopenia | 1 month
Frequency of PLT counts <75×10⁹/L during the study period | 1 month
Incidence of dose modifications, delays, or discontinuations caused by thrombocytopenia | 1 month
Incidence of severe adverse events (SAEs) graded by CTCAE v5.0 criteria | 2 months